CLINICAL TRIAL: NCT00097994
Title: Does Menopause Matter?
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Rachel Hess, MD, MS, University of Pittsburgh
Other Study IDs: AG0010; 1K23AG024254-01 (NIH); STRIDE
Record Dates: First submitted 2004-12-01; First posted 2004-12-02 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Menopause
Keywords: Menopause; Quality of Life; Health Services; Complementary Therapies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to follow a woman's progression through menopause in order to examine the effects on health related quality of life and use of health care resources, and to understand how women are using alternative therapies.

DETAILED DESCRIPTION:
Menopause affects every woman as she ages, yet every woman's experience is different. We are seeking to enroll 720 women from the University of Pittsburgh's Division of General Internal Medicine Outpatient practice (GIMO) at all stages of menopause (pre-, peri-, and post-menopausal), between 40 and 65 years old. They will be followed for 5 years as they progress through menopause.

Women will complete yearly questionnaires during their usual doctor's visit (or by phone or online if necessary) regarding general health, menopause and menopausal symptoms, health related quality of life, traditional and alternative therapy use, social support, and attitudes towards menopause and aging.

We will combine this information with information from women's medical charts to look at how menopause and health related quality of life impact the use of health care resources. Additionally, some women may be asked about the use of health care resources, such as doctor's visits, hospitalizations and lab tests.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 40-65
* Patients in the University of Pittsburgh General Internal Medicine Oakland Practice
* Able to complete the Functional Assessment Screening Tablet (a touch-screen survey)

Exclusion Criteria:

* Refusal to participate

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women from the University of Pittsburgh's Division of General Internal Medicine Outpatient practice (GIMO)
Sampling Method: Non-Probability Sample
Enrollment: 732 (Actual)
Dates: Start 2004-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life Score | Baseline survey
  The average enrollment scores of the dependent variable HRQOL [the physical and mental component summaries (PCS and MCS) of the SF-36] will be compared among women at different stages of menopause using ANOVA. If the HRQOL scores are not normally distributed on the original scale, a transformation is necessary. We will examine the association between both the baseline presence and severity of symptoms (0-4) and HRQOL using regression techniques. The association between the use of HT (yes/no) and HRQOL will be analyzed by ANOVA. The association between the use of CAM and HRQOL will be analyzed by ANOVA. The association between attitudes towards menopause and HRQOL will be analyzed by linear regression. Confounders, including age, comorbid medical conditions, and social support, will be included in the models. A final model examining the impact of all factors on HRQOL will be created using stepwise linear regression.

SECONDARY OUTCOMES:
Menopause Management | Menopausal Status Schema designed from STRAW and SWAN At least yearly Study Questions Menopausal Symptoms Vaginal dryness and hot flashes At least yearly Study Questions HRQOL SF-36 At least yearly CIF Social Support ISEL Yearly Study Questions Attitudes
  We will record all methods used by women in the cohort to manage menopause. Methods will be categorized as use of: no method, HT, and CAM. A frequency table will quantify use of each method as well as type of CAM. We will analyze the relationship between both menopausal symptoms and attitudes towards menopause and methods used by Chi-square or contingency table tests.

OTHER OUTCOMES:
Relationship between HSU and our independent variables, HRQOL and menopausal stage at assessment. | Physician visits Hospitalizations Prescriptions With each HRQOL assessment Electronic Medical Record (MARS) abstraction as well as subject self-report Intrusiveness of Menopausal Symptoms Year 2 assessment and yearly Study Questions Sleep
  Using regression analysis techniques, we will examine the relationship between HSU and our independent variables, HRQOL and menopausal stage at assessment. The model will also adjust for confounders such as age and the number and type of comorbidities at the time of analysis. Because all women in the study cohort will have utilization data for at least one physician visit, we will use a linear regression model. If cost data are not normally distributed, we will apply appropriate transformations.
  We will calculate the concordance correlation coefficient to investigate correlation between HSU data extracted from MARS and that obtained by direct patient interview to uncover under-reporting in the MARS database.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Hess, MD, MSc, Principal Investigator — UPMC General Internal Medicine-Oakland
Locations (1):
- UPMC General Internal Medicine Oakland, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Hlatky MA, Boothroyd D, Vittinghoff E, Sharp P, Whooley MA; Heart and Estrogen/Progestin Replacement Study (HERS) Research Group. Quality-of-life and depressive symptoms in postmenopausal women after receiving hormone therapy: results from the Heart and Estrogen/Progestin Replacement Study (HERS) trial. JAMA. 2002 Feb 6;287(5):591-7. doi: 10.1001/jama.287.5.591. PMID 11829697
- [Background] Avis NE, Ory M, Matthews KA, Schocken M, Bromberger J, Colvin A. Health-related quality of life in a multiethnic sample of middle-aged women: Study of Women's Health Across the Nation (SWAN). Med Care. 2003 Nov;41(11):1262-76. doi: 10.1097/01.MLR.0000093479.39115.AF. PMID 14583689
- [Background] Gambacciani M, Ciaponi M, Cappagli B, Monteleone P, Benussi C, Bevilacqua G, Genazzani AR. Effects of low-dose, continuous combined estradiol and noretisterone acetate on menopausal quality of life in early postmenopausal women. Maturitas. 2003 Feb 25;44(2):157-63. doi: 10.1016/s0378-5122(02)00327-4. PMID 12590012
- [Background] Albertazzi P, Purdie D. The nature and utility of the phytoestrogens: a review of the evidence. Maturitas. 2002 Jul 25;42(3):173-85. doi: 10.1016/s0378-5122(02)00024-5. PMID 12161041
- [Derived] Thomas S, Ness RB, Thurston RC, Matthews K, Chang CC, Hess R. Racial differences in perception of healthy body weight in midlife women: results from the Do Stage Transitions Result in Detectable Effects study. Menopause. 2013 Mar;20(3):269-73. doi: 10.1097/GME.0b013e31826e7574. PMID 23435023